CLINICAL TRIAL: NCT06907849
Title: PET/CT Imaging Of Subjects With Lumbar Spinal Stenosis Or Carpal Tunnel Syndrome Using Amyloid-Reactive Peptide 124I-Evuzamitide
Brief Title: 124I-Evuzamitide PET/CT Imaging In Patients With Lumbar Spinal Stenosis and Carpal Tunnel Syndrome
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Attralus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UTGSM-172768-101
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spinal Stenosis; Carpal Tunnel Syndrome (CTS); Cardiac Amyloidosis
Keywords: iodine-124-evuzamitide; PET Imaging; Amyloidosis; Spinal Stenosis; Carpal Tunnel Syndrome; p5+14
MeSH Terms: conditions — Spinal Stenosis; Carpal Tunnel Syndrome; Amyloid Neuropathies, Familial; Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biodistribution (Experimental): Participants will be administered ~1 mCi of 124I-evuzamitide (up to 1 mg of peptide) by IV push at a proposed rate of ~1 mL per 5 seconds. Three hours after injection, a PET/CT image acquisition from shoulder to thigh as well as a 10 min static PET image of the heart will be performed.
  Interventions: Drug: 124I-evuzamitide

INTERVENTIONS:
Drug: 124I-evuzamitide — 124I-evuzamitide is an iodine-124 (124I) labeled 45 L-amino acid peptide (also known as p5+14) suitable for single dose PET/CT imaging. The peptide binds many forms of amyloid through multivalent electrostatic interactions with the amyloid fibril and with the ubiquitous amyloid-associated hypersulfated heparan sulfate proteoglycans.
  Other Names: AT-01

SUMMARY:
This clinical trial will use the amyloid-binding radiotracer, 124I-evuzamitide, to potentially detect amyloid, in the heart and elsewhere, in patients who have a history of lumbar spinal stenosis and/or carpal tunnel syndrome.

DETAILED DESCRIPTION:
This is a single center, open label, pilot study using an amyloid-reactive peptide labeled with iodine-124 (124I-evuzamitide) and PET/CT imaging to detect the presence of cardiac and extracardiac amyloid in patients who have undergone surgical intervention for lumbar spinal stenosis (LSS) or carpal tunnel syndrome (CTS) and who have amyloid-positive connective tissue [ligamentum flavum (LF) in LSS patients or tenosynovium in CTS patients] assessed at the time of the corrective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 60 years of age.
* Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.
* Must have a Congo red positive ligamentum flavum or tenosynovial specimen analysis after laminectomy or carpal tunnel release surgery that is visually categorized as either "extensive" amyloid load or "mild/moderate" amyloid load by an experienced reviewer.
* Those with mild/moderate amyloid load in the connective tissue who also have a history of at least one other orthopedic clinical manifestation, including, but not limited to, carpal tunnel syndrome, lumbar spinal stenosis, trigger finger, biceps tendon rupture, and shoulder/hip/knee arthroplasty.
* Females must be non-pregnant and non-lactating.

Exclusion Criteria:

* Subjects on dialysis.
* Subjects with a confirmed diagnosis of systemic amyloidosis, other than musculoskeletal tissue.
* Inability or unwillingness to comply with the study requirements.
* Subjects taking heparin, or heparin derivatives (e.g. low molecular weight heparins) for anticoagulation.
* Inability to lie still for ~40 minutes on the PET/CT scanner.
* History of iodine (potassium iodide) allergy.
* Other reason that would make the subject inappropriate for entry into this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Detection of cardiac amyloidosis using 124I-evuzamitide PET/CT imaging | From enrollment to the end of study is 8 days.
  Cardiac PET/CT images will be classified as either positive or negative for 124I-evuzamitide uptake based on visual interpretation.

SECONDARY OUTCOMES:
Measure uptake of 124I-evuzamitide radioactivity in the heart and compare to biomarkers | From enrollment to the end of study is 8 days.
  Measure cardiac 124I-evuzamitide uptake and compare to contemporaneous transthoracic echocardiographic parameters, serum NT-proBNP, and high sensitivity troponin T levels
Measure uptake of 124I-evuzamitide radioactivity in the heart and compare to amyloid load in connective tissue | From enrollment to the end of study is 8 days.
  Measure cardiac 124I-evuzamitide uptake and compare to the reported amyloid load, based on Congo red staining, in connective tissue (obtained from LSS or CTS surgery)
Detection of extracardiac amyloid using 124I-evuzamitide PET/CT imaging | From enrollment to the end of study is 8 days.
  Visual examination of extracardiac 124I-evuzamitide uptake in the PET/CT images

CONTACTS AND LOCATIONS:
Overall Officials: Emily B. Martin, PhD, Principal Investigator — University of Tennessee Graduate School of Medicine
Locations (1):
- University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wall JS, Martin EB, Lands R, Ramchandren R, Stuckey A, Heidel RE, Whittle B, Powell D, Richey T, Williams AD, Foster JS, Guthrie S, Kennel SJ. Cardiac Amyloid Detection by PET/CT Imaging of Iodine (124I) Evuzamitide (124I-p5+14): A Phase 1/2 Study. JACC Cardiovasc Imaging. 2023 Nov;16(11):1433-1448. doi: 10.1016/j.jcmg.2023.08.009. PMID 37940323